CLINICAL TRIAL: NCT04569565
Title: Prospective Evaluation of PleurX Drain for Treatment of Cirrhotic Refractory Ascites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00055611
Record Dates: First submitted 2020-09-22; First posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Ascites Hepatic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PleurX catheter intervention (Experimental): Participants will undergo placement and follow up monitoring of PleurX catheter.
  Interventions: Device: PleurX catheter

INTERVENTIONS:
Device: PleurX catheter — Placement of PleurX catheter for refractory cirrhotic ascites, with follow up monitoring

SUMMARY:
Refractory ascites (fluid build up in the abdomen that can not bet managed by medications) occurs in at least 10% of patients with end stage liver disease (cirrhosis). Two major options for management include large volume paracentesis (LVP)-drainage with a needle through the abdominal wall) and placement of a transjugular intrahepatic portosystemic shunt (TIPS)-re-directs blood flow across the cirrhotic liver), Not all patients are candidates for TIPS or transplant, are left with LVP as the only long-term treatment option. Patients listed for transplant require LVP while they wait for transplant.

LVP can cause pain, bleeding, leakage from the drain site and frequent hospital visits which result in health care cost as well as patient and caregiver fatigue. In between the drains, living with ascites can negatively affect quality of life because of discomfort and limitations. Patients with ascites are more malnourished than those without.

Specialized drains tunnelled under the skin, are used in patents with ascites due to cancer (malignant). There are not many studies evaluating these drains in patients with cirrhosis, One of the reasons for the lack of studies is the potential for infection. As opposed to malignant ascites, cirrhotic ascites generally has a low protein content, a risk factor for development of spontaneous bacterial peritonitis (SBP). From available studies, infection rates in cirrhotic patients with tunnelled drains who are not on antibiotics are estimated at 10% (4/40). Infection rates on antibiotic prophylaxis would be expected to be lower.

This pilot study includes the evaluation of indwelling tunnelled PleurX catheters as an alternative option. The hypothesis is that with careful monitoring of kidney function and prevention of infection with antibiotics, PleurX catheters will be safe, cost-effective and improve quality of life and nutritional status compared to the standard of care.

DETAILED DESCRIPTION:
Ascites not manageable by diuretic therapy occurs in at least 10% of patients with cirrhosis. Two major options for management include intermittent large volume paracentesis (LVP) and placement of a transjugular intrahepatic portosystemic shunt (TIPS). Unfortunately, not all patients are candidates for TIPS. Those unable to receive TIPS or transplant are left with LVP as the only long-term treatment option. Non-TIPS candidates who are listed for transplant require LVP as a bridge to transplant.

LVP is performed by inserting a non-tunnelled drain, removing ascites fluid via, replacing ascites fluid losses >5 litres(L) with albumin, removing the drain. It can be associated with pain, bleeding, leakage from the site and frequent hospital visits. In between the drains, living with ascites can negatively affect quality of life, particularly the physical discomfort and limitation component scales. In addition, patients with tense ascites have lower protein intake and are more malnourished than those without. Fluid removal improves gastric accommodation.

Indwelling ascites drains are routinely used in patents with malignant ascites. Data evaluating indwelling drains in patients with cirrhosis is limited. One of the reasons that this may not have been explored as a therapeutic option is the potential for infection. As opposed to malignant ascites, cirrhotic ascites generally has a low protein content, a known risk factor for development of spontaneous bacterial peritonitis (SBP). From available data, infection rates in cirrhotic patients with tunnelled drains, not on antibiotic prophylaxis are estimated at 10%. Infection rates on antibiotic prophylaxis would be expected to be lower, but this remains unstudied. Other concerns particular to the patient with cirrhosis are renal dysfunction and acute kidney injury. Limitation of the amount of ascites that is drained to <5L per time and infusion of albumin 8grams(g)/L removed for amounts drained >5L has shown benefit in preventing post paracentesis circulatory and renal dysfunction.

Therefore, as some patients with cirrhosis will be left with intermittent LVP as their only option for management, and as this therapy has implications for quality of life (QOL), worsening nutritional status and cost, we propose an evaluation of an indwelling tunnelled PleurX catheter as an alternative therapeutic option. In this prospective uncontrolled pilot study, the hypothesis is that use of indwelling drains with careful monitoring of renal function and prophylaxis with antibiotics, will be safe, cost-effective and improve quality of life and nutritional status compared to the standard of care.

METHODS:

Study design: Prospective uncontrolled interventional pilot study of 12 patients followed for 3 months.

Recruitment: Patients will be recruited from Hepatology departments at the University of Alberta hospital (UAH) and Royal Alexandra hospital (RAH) in Edmonton. All Hepatologists at these sites will be informed of the protocol. If a patient meets inclusion and exclusion criteria and is interested in hearing more about the study, the Hepatologist can contact the study personnel. Patients will be made aware that their decision to participate in the study will not influence their medical care.

Study Intervention:

PleurX drain insertion by interventional radiologist

Outpatient drainage protocol:

Ascites fluid drainage performed at participant's home via home care nurse 1-3 times per week (maximum 3L- with each drain) for 3months. PleurX drain bottles will be used instead of urinary drainage bags

Safety Measures:

Home care nurses are trained in the use of PleurX drains. Patients will be taught and given information about complication monitoring.

Albumin infusion at 1g/kilogram(kg) as an outpatient when: the serum creatinine increases from baseline >26umol/L or by 1.5-2 times (Stage 1 Acute Kidney Injury), or the patient has clinical signs of hypovolemia Spontaneous bacterial peritonitis (SBP) prophylaxis with Norfloxacin 400mg daily Patient counselling on avoidance of non-steroidal anti-inflammatory drugs (NSAIDs), aminoglycosides, radiologic contrast, angiotensin converting enzyme (ACE) inhibitors, angiotensin II antagonists, angiotensin receptor blockers (ARBs) where possible

PROCEDURE & DATA COLLECTION:

Pre-Intervention (2 weeks prior to drain placement)

Continued standard of care LVP with albumin replacement, and recording of procedure related complications (shunt misplacement, insertion bleeding, pain-10 point scale) Pt to complete three-day food record (including 1 day pre-paracentesis, day of paracentesis, and 1 day post paracentesis), as well as Council on Nutrition appetite questionnaire (CNAQ, score range 8-40 where a lower score indicates more problems with appetite).

Nutritional assessment: Weight (kilograms), height (centimeters), calorie (kilocalories) and protein (grams) intake, mid-arm muscle circumference(centimeters), hand-grip strength by Jamar hand-grip dynamometer (kilograms) Labs pre-LVP including: urine electrolytes, serum complete blood cell (CBC) and differential, prothrombin time(PT), creatinine(Cr), electrolytes, alanine transaminase (ALT), aspartate transaminase (AST), Bilirubin, albumin, rennin, aldosterone

Quality of life and symptom questionnaires pre and post paracentesis: Chronic Liver Disease Questionnaire (CLDQ). The CLDQ includes 29 symptom questions, scored on a likert scale of 1-7 (where 1 is all of the time and 7 is none of time), and divided into 6 domains: fatigue, activity, emotional function, abdominal symptoms, systemic symptoms, and worry). Edmonton Symptom Assessment System-revised version (ESAS-R). The ESAS-R includes 10 symptoms (9 pre-determined and 1 'other' free text scale), scored on a likert scale 0-10 (where 0 is 'No' and 10 is 'Worst possible'). Ascites Symptom Inventory-7 (ASI-7). The ASI-7 includes 7 symptom questions, scored on a likert scale of 0-4 where 0 is 'does not apply at all' and 4 is 'very strongly applies'.

History and physical examination: Demographics, Past Medical History, Medications, History of prior ascites fluid infections, other infections, and antibiotic use in the last 6 months, Liver disease severity-model for end stage liver disease (MELD, score range 6-40, where a higher score indicates higher mortality risk ) score & Child Pugh score (score range 5-15, where a higher score indicates worse liver function), Resting blood pressure.

Day 1-90 (Day 1=drain placement day)

Adverse event monitoring and patient follow-up:

Pre-drain insertion abdominal wall ultrasound by the interventional radiologist who will be inserting the drain Drain placement associated safety outcomes will be recorded including: shunt misplacement, insertion bleeding, pain (10 point scale where 0 is 'no pain' and 10 is 'worst possible pain') Home care nurse visit assessment with each drain: vital signs, documentation of drain function, appearance, fluid drainage, fluid volume, fluid appearance, drain site description, patient symptoms.

Nurses will be asked to contact study personnel in the event of adverse outcomes or new patient symptoms Phone call to patient weekly and in person assessment monthly by primary investigator (PI): quality of life and symptom questionnaires-CLDQ, ESAS-R, ASI-7, changes in cognitive status, medication reassessment, documentation of hospitalizations, and Child Pugh/MELD calculation at monthly visit.

Monthly Nutritional assessment by dietitian-Weight, height, calorie and protein intake via 3-day food record (completed 1 day pre-drain, 1 day of a drain, and 1 day after a drain), mid-arm muscle circumference, hand-grip strength by the Jamar hand-grip dynamometer, CNAQ appetite screening tool

Diagnostic fluid analysis and septic work up if symptoms of SBP (abdominal pain, fever, elevated white blood cell count (WBC), sudden onset renal dysfunction or hepatic encephalopathy). Drain removal if SBP diagnosed using standard criteria (ascites fluid polymorphonuclear cell count ≥ 250 cells/millimetre3). Any removed drains with have the drain tip sent for culture and sensitivity

Labs: Weekly ascites fluid analysis for protein, cell count and diff, culture and sensitivity Weekly CBC and differential, PT, Cr, electrolytes, ALT, AST, Bilirubin, albumin via home collections or community based lab. Urine electrolytes, Plasma renin & aldosterone monthly

STUDY EXTENSION OPTION

At 90 days, all patients that choose to continue with fluid drainage as per the study protocol, will be offered the option to continue contributing data to the study for the duration of time they have the drain inserted, or until they no longer wish to participate. Patients will be made aware that their decision to continue to participate in the study will not influence their medical care.

For patients that agree to continue participating, the initial protocol for drain frequency, volume, care, and safety measures will be followed. Data will be collected, including:

Every 4 weeks by PI or designate: quality of life and symptom questionnaires-CLDQ, ESAS-R, ASI-7, changes in cognitive status, medication reassessment, documentation of hospitalizations, and Child Pugh/MELD calculation, vital signs, documentation of drain function, appearance, drain site description, patient symptoms. Patients will be asked to bring in their home drain volume records for review at these visits. Nutritional assessment by dietitian-Weight, height, calorie and protein intake via 3-day food record (completed 1 day pre-drain, 1 day of a drain, and 1 day after a drain), mid-arm muscle circumference, hand-grip strength by the Jamar hand-grip dynamometer, CNAQ appetite screening tool.

Diagnostic fluid analysis and septic work up if symptoms of SBP (abdominal pain, fever, elevated WBC, sudden onset renal dysfunction or hepatic encephalopathy) Drain removal if SBP diagnosed using standard criteria (ascites fluid polymorphonuclear cell count ≥ 250 cells/mm3). Any removed drains with have the drain tip sent for culture and sensitivity.

Labs: Every 1-2 weeks-ascites fluid analysis for protein, cell count and diff, culture and sensitivity. Blood for CBC and differential, PT, Cr, electrolytes, AST, Bilirubin, albumin Every 4 weeks- blood rennin and aldosterone. Urine electrolytes.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis (based on imaging, liver function test abnormalities, biopsy, or portal hypertension associated complications)
* Refractory or resistant ascites
* Not a candidate for TIPS (hospital admissions for encephalopathy, Model for End Stage Liver Disease (MELD) ≥18, diastolic dysfunction (defined as E/A ratio <1 on echocardiogram), patient declined, advanced age, renal disease)
* Requiring large volume paracentesis ≥twice/month

Exclusion Criteria:

* Malignant ascites due to peritoneal carcinomatosis (requires positive fluid cytology)
* Patient unwilling to let home care staff enter home
* Patient unwilling to have intravenous albumin
* Patient unwilling to have drain placed
* Patients post liver transplant
* multi-loculated ascites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-05-18 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Ascites Symptom Inventory (ASI-7) | Change from baseline to 6 months
  Includes 7 symptom questions, scored on a Likert scale of 0-4 where 0 is 'does not apply at all' and 4 is 'very strongly applies'

SECONDARY OUTCOMES:
Model for End Stage Liver Disease - Sodium (MELD-Na) score | Change from baseline to 6 months
  Score range 6-40, where a higher score indicates higher mortality risk
Level of serum creatinine | Change from baseline to 6 months
  Physiological parameter measure un umol/L
Council on Nutrition Appetite Questionnaire (CNAQ) | Change from baseline to 6 months
  Includes 8 questions where total score range is 8-40. A lower score indicates more problems with appetite
Level of serum albumin | Change from baseline to 6 months
  Physiological parameter expressed in g/dL
Cost of care | Change from baseline to 6 months
  Expressed in Canadian dollars (CAD)
Chronic Liver Disease Questionnaire (CLDQ) | Change from baseline to 6 months
  Includes 29 symptom questions, scored on a Likert scale of 1-7 (where 1 is all of the time and 7 is none of time), and divided into 6 domains: fatigue, activity, emotional function, abdominal symptoms, systemic symptoms, and worry)
Edmonton Symptom Assessment System-revised version (ESAS-R) | Change from baseline to 6 months
  Includes 10 symptoms (9 pre-determined and 1 'other' free text scale), scored on a Likert scale 0-10 (where 0 is 'No' and 10 is 'Worst possible')
Total calorie and protein intake | Change from baseline to 6 months
  Total food and drink intake is recorded for 3 days. Total calorie and protein (grams) intake are then calculated based on reported intake.
Visual Analog Pain scale | Change from baseline to 6 months
  Likert scale 0-10, where 0 is no pain and 10 is worst possible pain.
Child Pugh score | Change from baseline to 6 months
  Score range 5-15, where a higher score indicates worse liver function

CONTACTS AND LOCATIONS:
Overall Officials: Puneeta Tandon, Principal Investigator — University of Alberta; Juan G Abraldes, Principal Investigator — University of Alberta

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with other researchers

REFERENCES:
- [Background] Po CL, Bloom E, Mischler L, Raja RM. Home ascites drainage using a permanent Tenckhoff catheter. Adv Perit Dial. 1996;12:235-6. PMID 8865911
- [Background] Savin MA, Kirsch MJ, Romano WJ, Wang SK, Arpasi PJ, Mazon CD. Peritoneal ports for treatment of intractable ascites. J Vasc Interv Radiol. 2005 Mar;16(3):363-8. doi: 10.1097/01.RVI.0000147082.05392.2B. PMID 15758132
- [Background] Nadir A, Van Thiel DH. Frequency of peritoneal infections among patients undergoing continuous paracentesis with an indwelling catheter. J Ayub Med Coll Abbottabad. 2010 Jan-Mar;22(1):37-41. PMID 21409900
- [Background] Reinglas J, Amjadi K, Petrcich B, Momoli F, Shaw-Stiffel T. The Palliative Management of Refractory Cirrhotic Ascites Using the PleurX ((c)) Catheter. Can J Gastroenterol Hepatol. 2016;2016:4680543. doi: 10.1155/2016/4680543. Epub 2016 Jun 5. PMID 27446840
- [Background] Reisfield GM, Wilson GR. Management of intractable, cirrhotic ascites with an indwelling drainage catheter. J Palliat Med. 2003 Oct;6(5):787-91. doi: 10.1089/109662103322515365. No abstract available. PMID 14622465
- [Background] Bellot P, Welker MW, Soriano G, von Schaewen M, Appenrodt B, Wiest R, Whittaker S, Tzonev R, Handshiev S, Verslype C, Moench C, Zeuzem S, Sauerbruch T, Guarner C, Schott E, Johnson N, Petrov A, Katzarov K, Nevens F, Zapater P, Such J. Automated low flow pump system for the treatment of refractory ascites: a multi-center safety and efficacy study. J Hepatol. 2013 May;58(5):922-7. doi: 10.1016/j.jhep.2012.12.020. Epub 2013 Jan 11. PMID 23318604
- [Background] European Association for the Study of the Liver. EASL clinical practice guidelines on the management of ascites, spontaneous bacterial peritonitis, and hepatorenal syndrome in cirrhosis. J Hepatol. 2010 Sep;53(3):397-417. doi: 10.1016/j.jhep.2010.05.004. Epub 2010 Jun 1. No abstract available. PMID 20633946
- [Background] Patel PA, Ernst FR, Gunnarsson CL. Evaluation of hospital complications and costs associated with using ultrasound guidance during abdominal paracentesis procedures. J Med Econ. 2012;15(1):1-7. doi: 10.3111/13696998.2011.628723. Epub 2011 Oct 19. PMID 22011070
- [Background] White J, Carolan-Rees G. PleurX peritoneal catheter drainage system for vacuum-assisted drainage of treatment-resistant, recurrent malignant ascites: a NICE Medical Technology Guidance. Appl Health Econ Health Policy. 2012 Sep 1;10(5):299-308. doi: 10.1007/BF03261864. PMID 22779402
- [Background] Arroyo V. A new method for therapeutic paracentesis: the automated low flow pump system. Comments in the context of the history of paracentesis. J Hepatol. 2013 May;58(5):850-2. doi: 10.1016/j.jhep.2013.01.037. Epub 2013 Feb 8. No abstract available. PMID 23395692
- [Background] Les I, Doval E, Flavia M, Jacas C, Cardenas G, Esteban R, Guardia J, Cordoba J. Quality of life in cirrhosis is related to potentially treatable factors. Eur J Gastroenterol Hepatol. 2010 Feb;22(2):221-7. doi: 10.1097/MEG.0b013e3283319975. PMID 19794311
- [Background] Sola E, Watson H, Graupera I, Turon F, Barreto R, Rodriguez E, Pavesi M, Arroyo V, Guevara M, Gines P. Factors related to quality of life in patients with cirrhosis and ascites: relevance of serum sodium concentration and leg edema. J Hepatol. 2012 Dec;57(6):1199-206. doi: 10.1016/j.jhep.2012.07.020. Epub 2012 Jul 20. PMID 22824819
- [Background] Campbell MS, Brensinger CM, Sanyal AJ, Gennings C, Wong F, Kowdley KV, McCashland T, Reddy KR. Quality of life in refractory ascites: transjugular intrahepatic portal-systemic shunting versus medical therapy. Hepatology. 2005 Sep;42(3):635-40. doi: 10.1002/hep.20840. PMID 16108073
- [Background] Saiz-Mendiguren R, Gomez-Ayechu M, Noguera JJ, Garcia-Lallana A, Marginet C, Cano D, Benito A. [Permanent tunneled drainage for malignant ascites: initial experience with the PleurX(R) catheter]. Radiologia. 2010 Nov-Dec;52(6):541-5. doi: 10.1016/j.rx.2010.06.005. Epub 2010 Sep 21. Spanish. PMID 20863540
- [Background] Tapping CR, Ling L, Razack A. PleurX drain use in the management of malignant ascites: safety, complications, long-term patency and factors predictive of success. Br J Radiol. 2012 May;85(1013):623-8. doi: 10.1259/bjr/24538524. Epub 2011 Mar 22. PMID 21427184
- [Background] Courtney A, Nemcek AA Jr, Rosenberg S, Tutton S, Darcy M, Gordon G. Prospective evaluation of the PleurX catheter when used to treat recurrent ascites associated with malignancy. J Vasc Interv Radiol. 2008 Dec;19(12):1723-31. doi: 10.1016/j.jvir.2008.09.002. Epub 2008 Oct 31. PMID 18951041
- [Background] Johnson TM, Overgard EB, Cohen AE, DiBaise JK. Nutrition assessment and management in advanced liver disease. Nutr Clin Pract. 2013 Feb;28(1):15-29. doi: 10.1177/0884533612469027. PMID 23319353
- [Background] Angermayr B, Cejna M, Karnel F, Gschwantler M, Koenig F, Pidlich J, Mendel H, Pichler L, Wichlas M, Kreil A, Schmid M, Ferlitsch A, Lipinski E, Brunner H, Lammer J, Ferenci P, Gangl A, Peck-Radosavljevic M. Child-Pugh versus MELD score in predicting survival in patients undergoing transjugular intrahepatic portosystemic shunt. Gut. 2003 Jun;52(6):879-85. doi: 10.1136/gut.52.6.879. PMID 12740346
- [Background] Riggio O, Angeloni S, Salvatori FM, De Santis A, Cerini F, Farcomeni A, Attili AF, Merli M. Incidence, natural history, and risk factors of hepatic encephalopathy after transjugular intrahepatic portosystemic shunt with polytetrafluoroethylene-covered stent grafts. Am J Gastroenterol. 2008 Nov;103(11):2738-46. doi: 10.1111/j.1572-0241.2008.02102.x. Epub 2008 Sep 4. PMID 18775022
- [Background] Cazzaniga M, Salerno F, Pagnozzi G, Dionigi E, Visentin S, Cirello I, Meregaglia D, Nicolini A. Diastolic dysfunction is associated with poor survival in patients with cirrhosis with transjugular intrahepatic portosystemic shunt. Gut. 2007 Jun;56(6):869-75. doi: 10.1136/gut.2006.102467. Epub 2006 Nov 29. PMID 17135305
- [Background] Van Waes L, Demeulenaere L. [Treatment of intractable ascites using continued puncture re-infusion. The Rhodiascit system]. Tijdschr Gastroenterol. 1973;16(6):396-409. No abstract available. Dutch. PMID 4782125
- [Background] Leveen HH, Christoudias G, Ip M, Luft R, Falk G, Grosberg S. Peritoneo-venous shunting for ascites. Ann Surg. 1974 Oct;180(4):580-91. doi: 10.1097/00000658-197410000-00023. PMID 4415019
- [Background] Mehta RL, Kellum JA, Shah SV, Molitoris BA, Ronco C, Warnock DG, Levin A; Acute Kidney Injury Network. Acute Kidney Injury Network: report of an initiative to improve outcomes in acute kidney injury. Crit Care. 2007;11(2):R31. doi: 10.1186/cc5713. PMID 17331245
- [Background] Garcia-Tsao G, Parikh CR, Viola A. Acute kidney injury in cirrhosis. Hepatology. 2008 Dec;48(6):2064-77. doi: 10.1002/hep.22605. PMID 19003880
- [Background] Llach J, Rimola A, Navasa M, Gines P, Salmeron JM, Gines A, Arroyo V, Rodes J. Incidence and predictive factors of first episode of spontaneous bacterial peritonitis in cirrhosis with ascites: relevance of ascitic fluid protein concentration. Hepatology. 1992 Sep;16(3):724-7. doi: 10.1002/hep.1840160318. PMID 1505916
- [Background] Gines A, Fernandez-Esparrach G, Monescillo A, Vila C, Domenech E, Abecasis R, Angeli P, Ruiz-Del-Arbol L, Planas R, Sola R, Gines P, Terg R, Inglada L, Vaque P, Salerno F, Vargas V, Clemente G, Quer JC, Jimenez W, Arroyo V, Rodes J. Randomized trial comparing albumin, dextran 70, and polygeline in cirrhotic patients with ascites treated by paracentesis. Gastroenterology. 1996 Oct;111(4):1002-10. doi: 10.1016/s0016-5085(96)70068-9. PMID 8831595
- [Background] Campillo B, Richardet JP, Scherman E, Bories PN. Evaluation of nutritional practice in hospitalized cirrhotic patients: results of a prospective study. Nutrition. 2003 Jun;19(6):515-21. doi: 10.1016/s0899-9007(02)01071-7. PMID 12781851
- [Background] Wilson MM, Thomas DR, Rubenstein LZ, Chibnall JT, Anderson S, Baxi A, Diebold MR, Morley JE. Appetite assessment: simple appetite questionnaire predicts weight loss in community-dwelling adults and nursing home residents. Am J Clin Nutr. 2005 Nov;82(5):1074-81. doi: 10.1093/ajcn/82.5.1074. PMID 16280441
- [Background] Younossi ZM, Guyatt G, Kiwi M, Boparai N, King D. Development of a disease specific questionnaire to measure health related quality of life in patients with chronic liver disease. Gut. 1999 Aug;45(2):295-300. doi: 10.1136/gut.45.2.295. PMID 10403745
- [Background] Watanabe SM, Nekolaichuk C, Beaumont C, Johnson L, Myers J, Strasser F. A multicenter study comparing two numerical versions of the Edmonton Symptom Assessment System in palliative care patients. J Pain Symptom Manage. 2011 Feb;41(2):456-68. doi: 10.1016/j.jpainsymman.2010.04.020. Epub 2010 Sep 15. PMID 20832987
- [Background] Runyon BA; AASLD. Introduction to the revised American Association for the Study of Liver Diseases Practice Guideline management of adult patients with ascites due to cirrhosis 2012. Hepatology. 2013 Apr;57(4):1651-3. doi: 10.1002/hep.26359. No abstract available. PMID 23463403